CLINICAL TRIAL: NCT04022408
Title: "To Study the Role of Liquid Based Cytology (LBC) for Diagnosis and Characterization of Biliopancreatic Tumor s Compared With Standard Cytology and On-site Evaluation: A Non-inferiority Trail".
Brief Title: To Study the Role of Liquid Based Cytology (LBC) for Diagnosis and Characterization of Biliopancreatic Tumor s Compared With Standard Cytology and On-site Evaluation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ILBS-Biliopancreatic Tumor-01
Record Dates: First submitted 2019-07-08; First posted 2019-07-17 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Pancreatobiliary-Type Carcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid based cytology (Experimental): .Liquid-based cytology (LBC), enables cells to be suspended in a monolayer. LBC makes better cytological assessment possible with improved sensitivity and specificity, since fixation is better and nuclear details are well preserved in the technique. Preneoplasticand neoplastic cells are not obscured by other cells, such as normal epithelial and inflammatory cells. LBC techniques are currently applied to cytological samples from several tissues or fluids. They include uterine cervix , endometrium, aspirates from breast , thyroid tumors, ascites and pleural effusion, and urine , LBC technology is suggested as an appropriate diagnostic method for metastatic tumors in cerebrospinal fluid .
  Interventions: Diagnostic Test: Liquid based cytology
- Conventional cytology (Active Comparator): It is a gold standard for histopathological diagnosis of pancreatobiliary malignancies till date
  Interventions: Diagnostic Test: Conventional cytology

INTERVENTIONS:
Diagnostic Test: Liquid based cytology — Liquid based cytology
  Arms: Liquid based cytology
Diagnostic Test: Conventional cytology — Conventional cytology
  Arms: Conventional cytology

SUMMARY:
Liquid Based Cytology is a method of preparing samples for examination in cytopathology.Liquid-based cytology (LBC), enables cells to be suspended in a monolayer. LBC makes better cytological assessment possible with improved sensitivity and specificity, since fixation is better and nuclear details are well preserved in the technique. Conventional cytology is gold standard for biliopancreatic malignancy examination. This method is operator depended and have high inter observer variation . On site evaluation increases the sensitivity of conventional cytology but requires the presence of pathologist at the time of sampling . Our study will compare LBC with conventional cytology ,If found to be non inferior will be great help in centre were on site evaluation cannot be carried out . It will further reduce the interobserver variation

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients (or guardian) undergoing EUS guided sampling of suspected pancreato-biliary tumors

Exclusion Criteria:

* Patients on anti-platelet agents(including aspirin).
* Patients with deranged coagulation parameters, defined by platelet counts <75,000/mm3 and/or INR >1.8

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of LBC for diagnosis of Bilio-pancreatic tumors, compared to cytology, on-site evaluation, and cell-block preparation. | 0 day

SECONDARY OUTCOMES:
Comparison of liquid based cytology versus conventional cytology in the diagnosis of tumor with size < 2 cm or > 2 cm | 0 day
Comparison of liquid based cytology versus conventional cytology in the diagnosis of tumor with respect to site of tumor (pancreas biliary tract or gall bladder). | 0 day

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India